CLINICAL TRIAL: NCT05487547
Title: Feasibility of IPL Combined With RF for Treatment of DED Due to MGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-VBU-NUERA-OPT-22-01
Record Dates: First submitted 2022-07-31; First posted 2022-08-04 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Dry Eye Disease; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study arm (Experimental): Subjects will receive 4 treatments at 2-weeks intervals. Each treatment will consist of IPL administered on the malar region, followed by RF administered around the eye, followed by Meibomian gland expression (MGX). Follow-up will be conducted at 4 weeks after the 4th treatment session.
  Interventions: Device: IPL_RF_MGX

INTERVENTIONS:
Device: IPL_RF_MGX — intense pulsed light followed by Radiofrequency followed by meibomian gland expression

SUMMARY:
The purpose of this single-arm pilot study is to evaluate the feasibility and safety of combination therapy of intense pulsed light (IPL) and (Radiofrequency) RF for treatment of Dry eye disease (DED) due to Meibomian gland dysfunction (MGD).

DETAILED DESCRIPTION:
In the past several years, a large number of studies have demonstrated that several sessions of IPL followed by MGX lead to a long-term reduction in signs and symptoms of DED due to MGD, however benefits for the patient are expected only after 2 or 3 sessions. On the other hand, several researchers reported that application of RF around the eyelids provide immediate relief of DED symptoms (unpublished observations: Dr. Chantel Garcia). The efficacy of RF for reduction of DED signs and symptoms was also demonstrated in two clinical studies and one animal model of obstructive MGD. Despite the small number of studies with RF, these preliminary results suggest that the combination of IPL, MGX and RF could provide immediate symptomatic relief together with long-term improvement of signs and symptoms of DED. In addition, combination therapy might be useful to increase the efficacy of monotherapy RF or monotherapy IPL.

The purpose of this single-arm pilot study is to evaluate the feasibility and safety of combination therapy of IPL and RF for treatment of DED due to MGD. As far as we know this is the first study of its kind. Results of this current study will be useful to choose the most effective outcome measures, to estimate the risk to benefit ratio, and to anticipate the effect size. In the future, such information will be essential for evaluating the merits of this approach, by designing a powered and randomized controlled study.

.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to read, understand and sign an IC form
* 22 or older
* Self-assessed symptoms are consistent with moderate to severe dry eye (OSDI score ≥ 23)
* Signs of MGD, as detected in biomicroscopy
* Modified Meibomian Gland Score (mMGS) > 12 in the lower eyelid of at least one eye
* Fitzpatrick skin type I-IV
* Subject is willing to comply with all study procedures

Exclusion Criteria:

* Fitzpatrick skin type V or VI
* Pacemaker
* Any metal implants above the neck, excluding dental implants
* Dry Eye due to Sjogren
* LASIK/SMILE surgery, within 1 year prior to screening
* RK surgery
* Other ocular surgery or eyelid surgery, within 3 months prior to screening
* Recent ocular trauma, within 3 months prior to screening
* Pre-cancerous lesions or skin cancer in the planned treatment area
* Severe active allergies, or other severe uncontrolled eye disorders affecting the ocular surface
* Uncontrolled infections or uncontrolled immunosuppressive diseases
* Legally blind in either eye worse than 20/200
* Ocular surface abnormality that may compromise corneal integrity in either eye (e.g., prior chemical burn, Epithelial Basement Membrane Dystrophy (EBMD)
* Eyelid abnormalities that affect lid function in either eye, including: entropion, ectropion, tumor, blepharospasm, Grading staining in the lower third secondary to lagophthalmos, severe trichiasis, and severe ptosis
* Within 3 months prior to screening, use of photosensitive medication and/or herbs that may cause sensitivity to 560-1200 nm light exposure, including: Isotretinoin, Tetracycline, Doxycycline, and St. John's Wort
* Active sun burn in the treatment area
* Moderate to severely compromised corneal health as assessed by corneal fluorescein staining
* Anterior chamber inflammation
* Corneal edema
* 4 weeks wash out of all prescription eye drops, excluding artificial lubricants
* No more than 75% loss of meibomian glands, as evaluated with meibography, in either lower eyelid
* Any non-prescription product for dry eye, within 1 month from the study, excluding artificial lubricants
* Any condition revealed whereby the investigator deems the subject inappropriate for this study

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
modified meibomian gland score (mMGS) | 4 weeks after the 4th treatment session
  15 meibomian glands along the lower lid (5 nasal + 5 central + 5 temporal) will be gently expressed with the dedicated expression forceps. Each gland will be scored 0 to 3, as follows: 0 = clear liquid meibum; 1 = cloudy liquid meibum; 2 = inspissated meibum; 3 = blocked). mMGS will be evaluated as the sum of scores for these 15 glands.

SECONDARY OUTCOMES:
OSDI | 4 weeks after the 4th treatment session
  Ocular Surface Disease Index questionnaire
Eyelid appearance | 4 weeks after the 4th treatment session
  Eyelid appearance will be assessed with biomicroscopy at the slit lamp. Five features of the eyelids will be scored: lid margin vascularity, eyelid thickness, loss of eyelashes, conjunctival injection, and plugging of meibomian gland orifices. Each feature will be scored using a 4 point grading system: 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
Number of expressible glands | 4 weeks after the 4th treatment session
  Glands along the upper and lower lids will be squeezed with a dedicated expression forceps. The number of glands expressing any meibum (clear liquid, cloudy liquid, or inspissated) will be counted, per each eyelid separately.
NIBUT | 4 weeks after the 4th treatment session
  The non-invasive breakup time (NIBUT) will be measured with the tear film analysis feature of the Antares system (CSO). The subject will be asked to maintain his/her eye open, without blinking, in front of a device that will project concentric Placido disks will be projected onto the ocular surface. Mire reflections of these placido disks will be monitored. The first occurrence of image distortion will
Meibography | 4 weeks after the 4th treatment session
  The study investigator will invert the eyelids of the subject, to expose the meibomian glands. After viewing the inverted eyelids with infra-red light illumination using the Antares system (CSO), an infra-red image of the meibomian glands will be captured cand saved. The Antares software will be use to calculate the area of meibomian gland loss

OTHER OUTCOMES:
Predominant quality of the meibum | 4 weeks after the 4th treatment session
  The predominant quality of the meibum represents the quality of the meibum expressed from the majority of the meibomian glands. This will be assessed using a 4 point grading system: 0 = clear liquid, 1 = cloud liquid, 2 = inspissated, and 3 = no expression
MMP-9 test | 4 weeks after the 4th treatment session
  Presence/Absence of MMP-9 in tear samples will be evaluated with the InflammaDry test (Pathogen Screening, Sarasota, FL).

CONTACTS AND LOCATIONS:
Overall Officials: James Chelnis, MD, Principal Investigator — Manhattan Face and Eye; Chantel Garcia, OD, Principal Investigator — Carolina Eye Doctors
Locations (2):
- United States (2):
  - Manhattan Face and Eye clinic, New York, New York
  - Carolina Eye Doctors, Harrisburg, North Carolina

IPD SHARING:
Plan to Share IPD: No
No plan